CLINICAL TRIAL: NCT03633331
Title: A Phase II Trial Assessing the Tolerability of Palbociclib in Combination With Letrozole or Fulvestrant in Patients Aged 70 and Older With Estrogen Receptor-Positive, HER2-Negative Metastatic Breast Cancer
Brief Title: Palbociclib and Letrozole or Fulvestrant in Treating Patients With Estrogen Receptor Positive, HER2 Negative Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A171601; NCI-2017-01596 (Registry Identifier: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2018-08-07; First posted 2018-08-16 (Actual); Results first posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Estrogen Receptor-positive Breast Cancer; HER2/Neu Negative; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: interventions — palbociclib; Letrozole; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (palbociclib, letrozole or fulvestrant) (Experimental): Patients receive palbociclib PO QD on days 1-21. Patients also receive letrozole PO QD on days 1-28 or fulvestrant IM on days 1 and 15 of course 1 and on day 1 of subsequent courses per MD discretion. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Palbociclib; Drug: Letrozole; Drug: Fulvestrant; Other: Questionnaire Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Palbociclib — Given PO
Drug: Letrozole — Given PO
Drug: Fulvestrant — Given IM
Other: Questionnaire Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies

SUMMARY:
This phase II trial studies the side effects and how well palbociclib and letrozole or fulvestrant works in treating patients aged 70 years and older with estrogen receptor positive, HER2 negative breast cancer that has spread to other places in the body. Palbociclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as letrozole or fulvestrant, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving palbociclib and letrozole or fulvestrant may work better in treating patients with breast cancer. The trial will explore factors other than chronologic age that can affect toxicity rates as identified using a cancer-specific geriatric assessment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the safety and tolerability (adverse event rate) of the combination of palbociclib and letrozole or fulvestrant in adults age 70 or older with estrogen receptor-positive, HER2-negative metastatic breast cancer.

SECONDARY OBJECTIVES:

I. To describe the full toxicity profile including all grade 2 and higher adverse events (per National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version [v.] 5.0), specifically estimating the rate of grade 2 and higher myelosuppression (neutropenia, leukopenia, thrombocytopenia, and anemia), neutropenic fever, gastrointestinal (GI) side effects (nausea, diarrhea, decreased appetite, vomiting, mucositis-oral), fatigue, neuropathy, and thromboembolism.

II. To describe rates of dose reductions, dose holds, and hospitalizations. III. To estimate median time to treatment failure, including progression free survival and overall survival.

IV. To estimate the rate of adherence to palbociclib, letrozole and fulvestrant.

V. To explore factors other than chronologic age that can affect toxicity rates as identified using a cancer-specific geriatric assessment.

VI. To describe the results of the Overall Treatment Utility (OTU). VII. To determine the degree of agreement between patient-reported adverse events (AEs) using Patient Reported Outcomes (PRO)-CTCAE measures and those reported using traditional collections for AEs.

VIII. To examine the association between sarcopenia and the development of toxicity and adverse events.

OUTLINE:

Patients receive palbociclib orally (PO) once daily (QD) on days 1-21. Patients also receive letrozole PO QD on days 1-28 or fulvestrant intramuscularly (IM) on days 1 and 15 of course 1 and on day 1 of subsequent courses per Doctor of Medicine (MD) discretion. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of disease: estrogen receptor positive and/or progesterone receptor (PR) positive, HER2 negative metastatic breast cancer; histologic confirmation is required
* Measurable disease or non-measurable disease
* Planning to begin palbociclib for metastatic disease; one prior line of endocrine therapy and/or chemotherapy for metastatic disease is allowed; patients may begin or have already begun endocrine therapy before they start palbociclib treatment, but no more than two weeks prior to registration
* No prior therapy with a CDK inhibitor
* Resolution of all acute toxic effects of prior therapy or surgical procedures to CTCAE grade =< 1 (except alopecia) or to baseline toxicities prior to previous therapy or surgical procedures, prior to registration
* No untreated brain metastases; patients with treated brain metastases must have completed treatment with steroids to be eligible
* No known interstitial lung disease
* No second malignancies other than non-melanoma skin cancers or cervical carcinoma in situ; however, patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for >= 3 years
* No active infection requiring treatment with antibiotics
* Patients must be able to swallow and retain oral medication
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Patients must be able to read and comprehend English or Spanish
* Absolute neutrophil count (ANC) >= 1500/mm^3 (1.5 x 10^9/L)
* Platelet count >= 100,000/mm^3 (100 x 10^9/L)
* Creatinine clearance >= 30 ml/min calculated using the Cockcroft-Gault formula
* Total serum bilirubin =< 1.5 upper limit of normal (ULN) (< 3 ULN if Gilbert's disease)
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) =< 3 x ULN (=< 5.0 x ULN if liver metastases present)
* Alkaline phosphatase =< 2.5 x ULN (=< 5 x ULN if bone or liver metastases present)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2024-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mina Sedrak, MD, MS, Study Chair — City of Hope Comprehensive Cancer Center
Locations (447):
- United States (447):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - City of Hope Corona, Corona, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope Mission Hills, Mission Hills, California
  - Saint Joseph Hospital - Orange, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope - Santa Clarita, Santa Clarita, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope Upland, Upland, California
  - City of Hope West Covina, West Covina, California
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - The Watson Clinic, Lakeland, Florida
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Hawaii Oncology Inc-POB I, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Savio, ‘Aiea, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - UM Saint Joseph Medical Center, Towson, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Steward Saint Elizabeth's Medical Center, Brighton, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - McLaren-Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians-Lansing, Lansing, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Maple Grove Medical Center, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Oakey, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - The Dana-Farber Cancer Institute at Londonderry, Londonderry, New Hampshire
  - AtlantiCare Health Park-Cape May Court House, Cape May Court House, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health Cancer Institute at Huntington, Greenlawn, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Hematology Oncology Associates of Central New York-Onondaga Hill, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Novant Health Oncology Specialists-Kernersville, Kernersville, North Carolina
  - Novant Health Oncology Specialists-Mount Airy, Mount Airy, North Carolina
  - CarolinaEast Medical Center, New Bern, North Carolina
  - CarolinaEast Oncology and Hematology Associates, New Bern, North Carolina
  - Novant Health Oncology Specialists-Statesville, Statesville, North Carolina
  - Novant Health Oncology Specialists-Davidson County, Thomasville, North Carolina
  - Novant Health Oncology Specialists-Wilkesboro, Wilkesboro, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - UPMC Pinnacle Harrisburg, Harrisburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Farmington Health Center, Farmington, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Centra Lynchburg Hematology-Oncology Clinic Inc, Lynchburg, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours DePaul Medical Center, Norfolk, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Bon Secours Health Center at Harbour View, Suffolk, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sedrak MS, Lee MK, Ji J, Satele DV, Freedman RA, Poorvu PD, O'Connor T, Williams GR, Hopkins JO, Muss HB, Cohen HJ, Partridge AH, Carey LA, Chow SL, Subbiah N, Le-Rademacher J, Jatoi A. Palbociclib in adults aged 70 years and older with advanced breast cancer: A phase 2 multicenter trial (Alliance A171601). J Geriatr Oncol. 2024 Jul;15(6):101813. doi: 10.1016/j.jgo.2024.101813. Epub 2024 Jun 8. PMID 38852379

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Palbociclib, Letrozole or Fulvestrant): Patients receive palbociclib PO QD on days 1-21. Patients also receive letrozole PO QD on days 1-28 or fulvestrant IM on days 1 and 15 of course 1 and on day 1 of subsequent courses per MD discretion. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Palbociclib: Given PO Letrozole: Given PO Fulvestrant: Given IM Questionnaire Administration: Ancillary studies>
  > Quality-of-Life Assessment: Ancillary studies
Period: Overall Study
Arm/Group | Treatment (Palbociclib, Letrozole or Fulvestrant)
Started | 93
Completed | 92
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Palbociclib, Letrozole or Fulvestrant)
Number analyzed (Participants) | 93
Age, Continuous [Median (Full Range); unit: years] | 74 [70 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 88
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 85
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: Defined as the proportion of patients with documentation of grade 3 - 5 toxicity (regardless of attribution using the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version [v.] 5.0 criteria). A 95% binomial confidence interval for single proportions will be constructed for the severe toxicity rate during treatment. Univariate relationships between the primary endpoint and various pre-treatment patient characteristics such as anemia, self-assessed functional status, or social support will be described via cross-tabulation and Fisher's exact testing. Exploratory logistic regression modeling, with limited generalizability due to the modest sample size, will be used to assess the relative contributions of these variables impact the likelihood of developing a severe toxicity during treatment. The strength of this association will be expressed in terms of an odds ratio and its associated 95% confidence interval.
Time Frame: 6 months
Population: patients meeting the eligibility criteria who have not withdrawn before treatment and have adverse event data available are considered evaluable for the primary endpoint.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Treatment (Palbociclib, Letrozole or Fulvestrant)
Number analyzed (Participants) | 90
proportion of patients | 0.756 [0.654 to 0.840]

2. Secondary Outcome: Incidence of Drug Toxicities - Measured by National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] v. 5.0
Description: Measured by National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] v. 5.0
Time Frame: Up to 1 year
Reporting Status: Not Posted, anticipated posting 2022-09

3. Secondary Outcome: Dose Reduction, Dose Hold, and Hospitalization Reasons
Description: A 95% binomial confidence interval for single proportions will be constructed for the percentage of patients that had at least one dose reduction, dose hold, or hospitalization within the first year of treatment.
Time Frame: Up to 1 year
Reporting Status: Not Posted, anticipated posting 2022-09

4. Secondary Outcome: Time to Treatment Failure (and Reason for Coming Off Study - Toxicity, Patient Preference, Progression)
Description: Distributions time to treatment failure will be estimated using Kaplan-Meier methodology. Treatment failure is defined as a severe adverse event, disease progression or patient refusal to continue assigned treatment. Any reason that treatment is discontinued to time to treatment failure and not censor patients will be included. The reason for treatment discontinuation will be captured.
Time Frame: Up to 5 years
Reporting Status: Not Posted

5. Secondary Outcome: Palbociclib Adherence Rate
Description: Patients to be included in the analysis cohort will be those patients who have taken one or more doses of the study treatment. Those patients will be considered adherent to study treatment. For each of the first 3 cycles, an estimate of the proportion of patients who meet the criteria for adherence and its corresponding 95% confidence interval will be determined.
Time Frame: Up to 12 weeks
Reporting Status: Not Posted, anticipated posting 2021-12

6. Secondary Outcome: Response Rate as Determined by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: The response rate is defined as the proportion of patients whose disease status met Response Evaluation Criteria in Solid Tumors (RECIST) criteria for complete response (CR) or partial response (PR) on 2 consecutive evaluations at least 8 weeks apart. A 95% binomial confidence interval for the response rate will be constructed.
Time Frame: Up to 1 year
Reporting Status: Not Posted, anticipated posting 2022-09

7. Secondary Outcome: Progression Free Survival (PFS)
Description: Distributions of progression free survival (PFS) times will be estimated using Kaplan-Meier methodology.
Time Frame: From start of treatment to the first of the following disease events: local/regional/distant recurrence, invasive contralateral breast disease, second primary or death due to any cause, assessed up to 5 years
Reporting Status: Not Posted, anticipated posting 2022-09

8. Secondary Outcome: Overall Survival (OS)
Description: Distributions of overall survival (OS) times will be estimated using Kaplan-Meier methodology.
Time Frame: Up to 5 years
Reporting Status: Not Posted

9. Secondary Outcome: Overall Treatment Utility (OTU) Results
Description: OTU is a novel composite endpoint developed by investigators of the FOCUS2 trial to assess the outcome of palliative chemotherapy. The patient will be given either an overall score of "good", "intermediate", or "poor". A 95% binomial confidence interval will be constructed for the percentage of patients that scored "good" on the OTU.
Time Frame: Up to 1 year
Reporting Status: Not Posted

10. Secondary Outcome: Sarcopenia Analysis
Description: Will examine variables associated with skeletal muscle loss during treatment and whether skeletal muscle loss during treatment is associated with the presence of grade 3-5 toxicity and adverse events. Sarcopenia will be treated as a binary variable using the Skeletal Muscle Index (SMI) (SMI < 41 cm^2/m^2 vs. SMI > 41 cm^2/m^2) and differences in grades chemotherapy toxicity and adverse events will be analyzed using two group t-tests and fisher's exact test. The number of patients with and without sarcopenia grouped by patients with or without grade 3+ Adverse Events (AE's) will be also be reported.
Time Frame: Up to 1 year
Reporting Status: Not Posted

11. Secondary Outcome: Quality of Life as Measured by the European Quality of Life Five Dimension Three Level Questionnaire (EQ-5D-3L)
Description: European Quality of Life Five Dimension Three Level Questionnaire (EQ-5D-3L) is comprised of 5 dimensions. Mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels, no problems, some problems, extreme problems. The EQ-5D-3L can be converted to a single summary index. The median and range of this total score will be reported.
Time Frame: Up to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment (Palbociclib, Letrozole or Fulvestrant)
All-Cause Mortality (participants affected / at risk) | 4/92
Serious Adverse Events (participants affected / at risk) | 35/92
Other Adverse Events (participants affected / at risk) | 92/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Palbociclib, Letrozole or Fulvestrant) (N=92)
Anemia (Blood and lymphatic system disorders) | 6 (19)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (2)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (8)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (5)
Mucositis oral (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 5 (7)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chills (General disorders) | 1 (2)
Death NOS (General disorders) | 1 (1)
Fatigue (General disorders) | 6 (10)
Fever (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (5)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (2)
Neutrophil count decreased (Investigations) | 10 (25)
Platelet count decreased (Investigations) | 3 (7)
White blood cell decreased (Investigations) | 8 (19)
Anorexia (Metabolism and nutrition disorders) | 1 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (4)
Stroke (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 1 (1)
Hot flashes (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 2 (3)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Palbociclib, Letrozole or Fulvestrant) (N=92)
Anemia (Blood and lymphatic system disorders) | 72 (549)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 3 (39)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (19)
Cardiac disorders - Other, specify (Cardiac disorders) | 3 (3)
Chest pain - cardiac (Cardiac disorders) | 3 (13)
Heart failure (Cardiac disorders) | 1 (20)
Mobitz (type) II atrioventricular block (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (4)
Hearing impaired (Ear and labyrinth disorders) | 2 (5)
Vertigo (Ear and labyrinth disorders) | 2 (5)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (44)
Blurred vision (Eye disorders) | 6 (54)
Cataract (Eye disorders) | 2 (17)
Dry eye (Eye disorders) | 3 (5)
Eye disorders - Other, specify (Eye disorders) | 3 (8)
Eye pain (Eye disorders) | 1 (2)
Watering eyes (Eye disorders) | 2 (22)
Abdominal distension (Gastrointestinal disorders) | 1 (6)
Abdominal pain (Gastrointestinal disorders) | 3 (9)
Bloating (Gastrointestinal disorders) | 2 (3)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 17 (63)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 40 (214)
Dry mouth (Gastrointestinal disorders) | 10 (53)
Dyspepsia (Gastrointestinal disorders) | 7 (39)
Dysphagia (Gastrointestinal disorders) | 4 (16)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 2 (10)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 9 (35)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 30 (135)
Nausea (Gastrointestinal disorders) | 40 (153)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 14 (25)
Chills (General disorders) | 6 (8)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 8 (32)
Fatigue (General disorders) | 78 (716)
Fever (General disorders) | 4 (5)
Flu like symptoms (General disorders) | 1 (1)
Gait disturbance (General disorders) | 2 (6)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1)
Injection site reaction (General disorders) | 3 (10)
Localized edema (General disorders) | 1 (7)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (9)
Pain (General disorders) | 19 (44)
Allergic reaction (Immune system disorders) | 1 (1)
Bone infection (Infections and infestations) | 1 (4)
Bronchial infection (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 3 (3)
Lip infection (Infections and infestations) | 1 (7)
Mucosal infection (Infections and infestations) | 1 (16)
Otitis externa (Infections and infestations) | 1 (4)
Otitis media (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (4)
Skin infection (Infections and infestations) | 2 (4)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 9 (10)
Urinary tract infection (Infections and infestations) | 7 (8)
Wound infection (Infections and infestations) | 1 (3)
Bruising (Injury, poisoning and procedural complications) | 5 (11)
Burn (Injury, poisoning and procedural complications) | 1 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 6 (6)
Fracture (Injury, poisoning and procedural complications) | 4 (4)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (2)
Alanine aminotransferase increased (Investigations) | 14 (49)
Alkaline phosphatase increased (Investigations) | 7 (29)
Aspartate aminotransferase increased (Investigations) | 12 (45)
Blood bilirubin increased (Investigations) | 1 (6)
Blood lactate dehydrogenase increased (Investigations) | 1 (14)
CD4 lymphocytes decreased (Investigations) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Creatinine increased (Investigations) | 20 (66)
Investigations - Other, specify (Investigations) | 4 (15)
Lymphocyte count decreased (Investigations) | 26 (96)
Neutrophil count decreased (Investigations) | 85 (885)
Platelet count decreased (Investigations) | 61 (379)
Weight gain (Investigations) | 1 (6)
Weight loss (Investigations) | 4 (10)
White blood cell decreased (Investigations) | 80 (897)
Anorexia (Metabolism and nutrition disorders) | 28 (96)
Dehydration (Metabolism and nutrition disorders) | 4 (5)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (6)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (15)
Hyperglycemia (Metabolism and nutrition disorders) | 22 (104)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (5)
Hyperlipidemia (Metabolism and nutrition disorders) | 2 (38)
Hypernatremia (Metabolism and nutrition disorders) | 2 (4)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (15)
Hypocalcemia (Metabolism and nutrition disorders) | 11 (25)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 6 (15)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (8)
Hyponatremia (Metabolism and nutrition disorders) | 7 (22)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (107)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 24 (129)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (31)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (6)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8 (19)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (5)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 3 (11)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (43)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (7)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (59)
Ataxia (Nervous system disorders) | 1 (7)
Cognitive disturbance (Nervous system disorders) | 1 (8)
Dizziness (Nervous system disorders) | 7 (12)
Dysgeusia (Nervous system disorders) | 8 (21)
Headache (Nervous system disorders) | 9 (16)
Memory impairment (Nervous system disorders) | 3 (15)
Nervous system disorders - Oth spec (Nervous system disorders) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (15)
Peripheral motor neuropathy (Nervous system disorders) | 2 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 36 (315)
Tremor (Nervous system disorders) | 3 (10)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (16)
Anxiety (Psychiatric disorders) | 7 (20)
Confusion (Psychiatric disorders) | 3 (6)
Depression (Psychiatric disorders) | 10 (15)
Insomnia (Psychiatric disorders) | 13 (72)
Irritability (Psychiatric disorders) | 1 (1)
Personality change (Psychiatric disorders) | 1 (3)
Chronic kidney disease (Renal and urinary disorders) | 3 (27)
Dysuria (painful urination) (Renal and urinary disorders) | 1 (5)
Glucosuria (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 4 (5)
Urinary frequency (Renal and urinary disorders) | 3 (15)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 2 (6)
Vaginal discharge (Reproductive system and breast disorders) | 1 (2)
Vaginal dryness (Reproductive system and breast disorders) | 1 (8)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (37)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (73)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 27 (102)
Dry skin (Skin and subcutaneous tissue disorders) | 14 (58)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (16)
Nail changes (Skin and subcutaneous tissue disorders) | 3 (8)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (18)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (13)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (8)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 2 (3)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 2 (3)
Hot flashes (Vascular disorders) | 17 (92)
Hypertension (Vascular disorders) | 21 (138)
Hypotension (Vascular disorders) | 3 (12)
Lymphedema (Vascular disorders) | 7 (37)
Thromboembolic event (Vascular disorders) | 5 (13)
Vascular disorders - Other, specify (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT03633331/Prot_SAP_ICF_000.pdf